CLINICAL TRIAL: NCT01868217
Title: A Retrospective Study to Investigate Prevalence of Capsular Bag Distention Syndrome and Its Influencing Factors
Status: Completed | Type: Observational
Sponsor: Evidence Based Cataract Study Group (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC-81100653
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Capsular Bag Distention Syndrome After Cataract Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
* To Investigate the Prevalence of Capsular Bag Distention Syndrome
* To Analyze Influencing Factors of Capsular Bag Distention Syndrome

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent uneventful phacoemulsification and posterior-chamber IOL implantation at the Eye and ENT Hospital of Fudan University, Xuhui, Shanghai, China, between November 2011 and December 2012

Exclusion Criteria:

* Patients with traumatic cataracts or zonular weakness were excluded from the study, as were eyes with intraoperative complications, such as a posterior capsule opening, radial tearing of the continuous curvilinear capsulorhexis (CCC), or inappropriate IOL implantation.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Who Underwent Cataract Surgery at Eye and ENT Hospital of Fudan University, Xuhui, Shanghai, China
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Dimension of the eyeball(mm) | 1 month